CLINICAL TRIAL: NCT03234504
Title: Development and Validation of a Novel Stereoacuity Test Using Head-mounted Display
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0507
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Normal Healthy Volunteers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal healthy volunteers

SUMMARY:
This prospective study investigated the validity and test-retest reliability of stereopsis test using head-mount display (HMD). Contour-based circles (crossed disparity: 1,960 to 195 arc of seconds(arc secs)) were generated as separate images on a high resolution phone display (Galaxy S7; Samsung, Suwon, Korea) using a HMD (Galaxy Gear VR; Samsung, Suwon, Korea). Two images were independently projected to each eye as graded circles with random dot background. While the position of the stimulus changed from among 3 possible locations, the subjects were instructed to select the circle with disparity by pressing the corresponding position on a keypad. The results of the new HMD stereotest were compared to those from standard Randot and TNO stereotests.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects who want or need to visual acuity test or to test for a prescription for glasses visited the hospital. 2. The Subjects' ages ranged from 19 to 60 years in the study.

Exclusion Criteria:

1. Ocular alignment was assessed with cover-uncover and alternate prism cover testing at distance and near. Significant exodeviation included exophoria was considered to be ≥6 prism diopters were excluded.
2. Subjects with a history of ocular surgery within 3 months of the study were excluded.
3. Foreigners or subjects who are unable to understand informed consent were excluded.
4. Subjects with a history of eye problems, including infection, inflammation, cataract, vitreous opacity or retinal diseases were excluded.
5. Subjects with corrected visual acuity of 20/32 in bad eye were excluded.
6. Subjects with significant refractive error considered to be ≥2.00 diopters of anisometropia were excluded.
7. A female who is pregnant, may be pregnant, or is lactating was excluded.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: normal healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Correlation between stereopsis with head mount display and stereopsis with Randot or TNO test | one visit
  Stereopsis results was expressed as arc sec. The association between log arc sec in stereopsis with HMD display and Randot or TNO test were evaluated. Using Bland Altman plot, the mean differences between two stereopsis results were compared.

SECONDARY OUTCOMES:
Test-retest variability of stereopsis using head mount display | one visit
  The intraclass coefficient was calculated between initial head mount display stereopsis result and retests.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No